CLINICAL TRIAL: NCT00449501
Title: A Two-week, Randomised, Double-blind Study Assessing the Onset of Effect Questionnaire Administered Pre-dose Versus Post-dose in Adult Subjects (≥ 18 Years) With Mild to Moderate Asthma, Receiving SYMBICORT® pMDI 80/4.5 μg x 2 Actuations Twice Daily or Budesonide HFA pMDI 80 μg x 2 Act. Twice Daily
Brief Title: A Two-week Study Assessing the Onset of Effect Questionnaire Administered Pre-dose Versus Post-dose in Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5896C00025
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Mild Asthma; Moderate Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Budesonide/formoterol pMDI
  Other Names: Symbicort
Drug: Budesonide HFA pMDI

SUMMARY:
The purpose of this study is to demonstrate whether subjects respond similarly to the Onset of Effect Questionnaire (OEQ) administered pre-dose versus post-dose, while receiving SYMBICORT® pMDI 80/4.5 μg x 2 actuations twice daily or budesonide HFA pMDI 80 μg x 2 actuations twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, > 18 years of age
* Mild to moderate asthma requiring treatment with an inhaled corticosteroid
* Diagnosis of asthma for at least 6 months

Exclusion Criteria:

* Subjects requiring treatment with systemic corticosteroids (e.g., oral, parenteral, ocular)
* Subjects with severe asthma, as judged by investigator
* Any significant disease or disorder that may jeopardize a subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine whether subjects respond similarly to the Onset of Effect Questionnaire items 2 and 5 when administered post-dose versus pre-dose and does that difference favour a bronchodilator treatment group over a non-bronchodilator treatment group

SECONDARY OUTCOMES:
To determine if there is an association between the immediate physiological response to medication and the responses to OEQ items 2 and 5 and to determine what subjects mean when they say they feel their asthma maintenance medication 'working right away

CONTACTS AND LOCATIONS:
Overall Officials: Tomas LG Andersson, MD, Study Director — AstraZenenca
Locations (46):
- United States (46):
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Los Angeles, California
  - Research Site, Palmdale, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Miami, Florida
  - Research Site, Avon, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Mandeville, Louisiana
  - Research Site, Wheaton, Maryland
  - Research Site, Bay City, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, McCook, Nebraska
  - Research Site, Scottsbluff, Nebraska
  - Research Site, Brick, New Jersey
  - Research Site, Princeton, New Jersey
  - Research Site, North Syracuse, New York
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Lake Oswego, Oregon
  - Research Site, Bensalem, Pennsylvania
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Watertown, South Dakota
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, Provo, Utah
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Leidy NK, Gutierrez B, Lampl K, Uryniak T, O'Brien CD. Can patients with asthma feel inhaler therapy working right away? Two clinical trials testing the effect of timing of assessment on patient perception. J Asthma. 2009 Dec;46(10):1006-12. doi: 10.3109/02770900903301260. PMID 19995138
- See also: Related Info — http://www.asthmaclinicaltrials.com